CLINICAL TRIAL: NCT01975181
Title: Cardiovascular Health Program Registry
Status: Terminated | Type: Observational
Why Stopped: No funding - program closure
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 372910
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular health; lifestyle modification; patient reported outcomes; risk assessment
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish a registry that uses observational study methods to collect uniform data (clinical, lifestyle and other) to evaluate specific outcomes and to enable research on patients at risk for cardiovascular disease (CVD).

This is a descriptive, observational registry study. All data for participants in the WRNMMC Integrative Cardiac Health Project (ICHP) Cardiovascular Health Program (CHP) will be entered into a single, secure information management system (IMS) for subjects at risk for CVD. At periodical intervals, the IMS will be queried to define the effect of an integrative therapeutic lifestyle change (TLC) program on CVD risk over time. This protocol outlines collection, storage, and handling of data, describes specific data elements and lays the foundation for future research questions.

DETAILED DESCRIPTION:
The CHP registry consists of uniform data to evaluate the outcomes of military beneficiaries at CVD risk. These uniform data include variables (clinical, lifestyle, traditional, non-traditional, objective and subjective) that are used to assess a CVD risk profile and the effects of TLC. All data are collected in the course of the clinical CHP.

Data are comprised of demographic information; past and intercurrent medical history including risk factors of CVD such as coronary artery disease (CAD), carotid disease, peripheral arterial disease, aortic aneurysm hypertension, diabetes and sleep apnea; smoking, alcohol and drug use history; family history of CVD and other chronic diseases; deployment history, injuries and occupational exposures; mental health history including PTSD, depression and anxiety; lifestyle information comprised of self-reported dietary patterns, exercise activities, stress levels, and sleep habits; physical examination including vital signs, body mass index, waist circumference and per cent body fat; laboratory data routinely requested by the CHP for risk assessment of all patients entering the program is comprised of total cholesterol, cholesterol fractions, fasting glucose, fasting insulin, hemoglobin A1C, highly sensitive C-reactive protein, and vitamin D levels; and CV diagnostic tests such as EKG, echocardiogram, cardiac stress testing; and sleep testing.

Data are measured at baseline (CHP enrollment), completion of onsite CHP (6 months) and after follow-up of the telephonic coaching phase (approximately 1 year). Data may also be collected annually for up to 5 years if available.

ELIGIBILITY:
Inclusion Criteria:

1. Any adult military, DEERS eligible, beneficiary who is participating in the CHP.
2. Subjects who present to the CHP for evaluation and participation may be self-referred or be referred by a provider.
3. Must have working email address and access to the internet.
4. Participants elect to enroll in order to learn about healthy lifestyle choices that can help prevent the development of cardiovascular disease.

Exclusion Criteria:

1. Less than 18 years of age.
2. Individuals unable or unwilling to participate or give informed consent will be excluded from registry enrollment.
3. Subjects who were part of the retrospective CHP cohort cannot be enrolled in the prospective study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 5000, male and female, adult military health care beneficiaries (active duty, dependents, and retired) who are at risk for CVD and who attend the CHP at WRNMMC will be asked to join the CHP registry. There will be no biased selection based on gender, age, racial or ethnic origin.
  A majority of participants are free of cardiovascular symptoms. Participants elect to enroll in order to learn about healthy lifestyle choices that can help prevent the development of cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Improvement in Cardiovascular Risk Score | 8 months
  A cardiovascular risk score is calculated using the Framingham Risk Score PLUS other factors including family history, body mass index, diastolic blood pressure, high sensitivity C-reactive protein, low-density lipoprotein, triglyceride and lipoprotein (a).

SECONDARY OUTCOMES:
Improvement in Dietary Score using the Rate-Your Plate Dietary Assessment Tool | 8 months
  Specific dietary behaviors are surveyed using the Rate-Your-Plate Dietary Assessment Tool with scores for each behavior ranging from 0 to 3. A high score indicates a health dietary behavior. All individual scores are added to calculate an overall score for healthy eating.
Improvement in Exercise | 8 months
  For exercise evaluation, questions concerning amounts of intentional exercise performed in at least 10 minute blocks will determine the activity levels individual patients are performing regularly.
Improvement in Perceived Stress Scale | 8 months
  Using the Perceived Stress Scale, subjects report on subjectively experienced stress levels over the several weeks prior to the measurement date.
Improvement in Pittsburgh Sleep Quality Index (PSQI) | 8 months
  Subjects complete the questionnaire (PSQI) to have a global assessment of their sleep quality for the time period including a month before the questionnaire completion.

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Villines, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Integrative Cardiac Health Project, Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Result] Eliasson AH, Kashani MD, Howard RS, Vernalis MN, Modlin RE; Integrative Cardiac Health Project Registry. Fatigued on Venus, sleepy on Mars-gender and racial differences in symptoms of sleep apnea. Sleep Breath. 2015 Mar;19(1):99-107. doi: 10.1007/s11325-014-0968-y. Epub 2014 Mar 15. PMID 24633816
- [Result] Kashani M, Eliasson AH, Walizer EM, Fuller CE, Engler RJ, Villines TC, Vernalis MN. Early Empowerment Strategies Boost Self-Efficacy to Improve Cardiovascular Health Behaviors. Glob J Health Sci. 2016 Sep 1;8(9):55119. doi: 10.5539/gjhs.v8n9p322. PMID 27157185